CLINICAL TRIAL: NCT02331771
Title: Can Donepezil Preserve Autobiographical Memory Post Electroconvulsive Therapy? A Randomized, Placebo-Controlled Trial
Brief Title: Donepezil Memory Preservation Post ECT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of sufficient enrollment
Sponsor: Porter Adventist Hospital (Other)
Responsible Party: Principal Investigator, Robin Wackernah, Pharmacist, Porter Adventist Hospital
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: PorterAH
Record Dates: First submitted 2014-12-31; First posted 2015-01-06 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Memory Impairment
MeSH Terms: conditions — Memory Disorders | interventions — Donepezil; Sucrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- donepezil (Active Comparator): Subjects will receive donepezil 5 mg before before they start ECT and continue the agent through the ECT procedures up to 4 weeks.
  Interventions: Drug: Donepezil
- Placebo (Placebo Comparator): Subjects will receive the placebo before they start ECT and continue the agent through the ECT procedures up to 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Donepezil — Donepezil 5 mg once daily 2 days before ECT and continuing through the last ECT procedure.
  Other Names: Aricept
  Arms: donepezil
Drug: Placebo — Placebo capsule once daily 2 days before ECT and continuing through the last ECT procedure.
  Other Names: Sucrose
  Arms: Placebo

SUMMARY:
This randomized, placebo-controlled trial will evaluate the use of donepezil compared to placebo to reduce the risk of memory impairment after electroconvulsive therapy (ECT).

DETAILED DESCRIPTION:
Electroconvulsive therapy (ECT) is a method used to treat a variety of psychiatric conditions. An electrical current is distributed throughout the brain (Lisanby 2007) inducing seizure activity in a controlled setting using neuromuscular blocking agents (Mirzakhani 2012) while the patient is under anesthesia (Deiner 2009). ECT is approved by the Food and Drug Administration (FDA) for the following conditions: unipolar and bipolar depression, manic and mixed states in bipolar disorder, schizophrenia, schizoaffective disorder, schizophreniform disorder and catatonia (FDA executive summary). ECT is often used after trials of psychotropic medications have failed (Kellner 2012).

Electroconvulsive therapy (ECT) is commonly associated with cognitive side effects that range from anterograde and retrograde amnesia to issues with executive function, attention and declines in information processing. Problems with autobiographical memory and recall for new information appear to be affected the most. In addition, data suggests that the loss of memory of autobiographical events may persist as long as six months. These issues may cause patient adherence problems and potential relapses into previous psychiatric conditions.

Donepezil is an acetylcholinesterase inhibitor indicated for Alzheimer's Dementia and has been shown to slow the progressive decline in cognition and memory in Alzheimer's Dementia. It is hypothesized that donepezil will help to preserve memory and minimize the decline in memory that is associated with the administration of ECT.

This study aims to determine if donepezil can minimize deficiencies in autobiographical memory 4-5 weeks after ECT treatment has been started.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depressive disorder, anxiety disorders, bipolar depression who are receiving right unilateral ECT will be included.

Exclusion Criteria:

* Patients with previous use of alcohol or illicit drugs within seven days of randomization will be excluded. Preexisting unstable cardiovascular disease including uncontrolled hypertension will be excluded. Patients with a documented allergy to donepezil will also be excluded. Patients with axis I disorders (eg. schizophrenia, schizoaffective disorder) other than major depressive disorder, anxiety disorders and/or bipolar depression will be excluded. Patients on anticoagulant therapy or chronic NSAID therapy will be excluded. Patients who are pregnant or wish to become pregnant within one year from trial enrollment will also be excluded. Patients who have received ECT within 6 months of enrollment will be excluded. Baseline Mini Mental State Examination (MMSE) < 24 will be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-09-24 (Actual); Primary Completion 2017-01-25 (Actual); Study Completion 2017-03-24 (Actual)

PRIMARY OUTCOMES:
Columbia University Autobiographical Memory Interview-Short Form (AMI-SF) | 4-5 weeks after first ECT treatment

SECONDARY OUTCOMES:
Short Term Memory Four-Word MemoryTask | 4-5 weeks after first ECT treatment

CONTACTS AND LOCATIONS:
Overall Officials: Robin Wackernah, Pharm.D., Principal Investigator — Pharmacist
Locations (1):
- Porter Adventist Hospital, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided